CLINICAL TRIAL: NCT06739447
Title: Implementing a Hospital-based Continuous Patient Monitoring System Using Consumer Wearable Devices in Ghana
Brief Title: Hospital Based Continuous Patient Monitoring System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Northwestern University (Other); University of Chicago (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); University of Ghana (Other); Loyola University (Other)
Responsible Party: Principal Investigator, Hassan Ghomrawi, Associate Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-300013798
Record Dates: First submitted 2024-11-22; First posted 2024-12-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Trauma; Appendectomy; Pediatric ALL; Vital Signs Monitoring
Keywords: Garmin Venu 3; pediatric appendectomy; trauma; vital sign monitoring
MeSH Terms: conditions — Wounds and Injuries; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Patients admitted to the Pediatric Trauma Unit in the Emergency Department and Pediatric Patients who have undergone an appendectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Consumer Wearable Device Measurement (Experimental): Consumer wearable devices (CWD)
  Interventions: Other: Consumer Wearable Device Vital Sign Measurement

INTERVENTIONS:
Other: Consumer Wearable Device Vital Sign Measurement — Consumer Wearable Devices such as the Fitbit, are durable devices that can provide vital sign data.

SUMMARY:
In Ghana, and many other low and middle income countries in Africa, manual vital signs monitoring is the prevalent mode of vital signs monitoring because continuous bedside monitors are non-functional. This lack of continuous vital signs monitoring may result in missed opportunities to catch physiologic deterioration.

The investigators propose to develop a dashboard that is based on the Garmin Venu 3, a consumer wearable device that reliably measures heart rate, SPO2, and respiratory rate, as an alternative to bedside monitors in hospitals in Ghana.

DETAILED DESCRIPTION:
Vital sign (VS) monitoring is a universal tool used to assess patients' basic physiologic status, primarily to detect physiologic deterioration indicative of clinically meaningful events. Physiologic deterioration occurs relatively commonly in trauma and postoperative patient populations. In most high-income countries (HIC), such patients are therefore monitored by automated, continuous, bedside VS systems, while, in many low-and middle-income countries (LMIC), manual, intermittent (from every 15 minutes to every 6 hours) VS monitoring is still widely employed.

The investigators propose to further refine and scale up a CONsumer-grade wearable monitoring System to improve Outcomes in Low resource settings (CONSOL) in Ghana. CONSOL is a CWD based platform, developed by the MPIs, that collects and displays in near real time, HR, RR, and SpO2, with snapshots of the past 1 minute, and 1, 4, and 24 hours, viewable on an tabet or smartphone. The investigators propose to evaluate the use of CONSOL for VS monitoring of (a) pediatric trauma patients in the Emergency Department (ED) and (b) pediatric postoperative appendicitis patients on a surgical unit, given higher risk of physiologic deterioration indicative of clinically meaningful events in these patient populations, and because pediatric patients are often more limited, than adults, in their ability to communicate about signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients presenting with traumatic injury
* Pediatric patients postoperative status after an appendectomy

Exclusion Criteria:

* Pediatric patients missing their upper limbs,
* Pediatric patients who cannot wear a Fitbit on their wrist for known allergies to rubber or those with traumatic or medical conditions that prevent them from being able to comfortably wear a Fitbit on either hand

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2029-11-30 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate with CONSOL compared to pre-CONSOL implementation | During the intervention (vital sign monitoring using the Garmin Venu 3)
  The investigators will implement CONSOL and record the abnormal vital signs indicative of clinically meaningful events in the CONSOL group. The investigators will then compare the number of abnormal vital signs detected in the CONSOL group to that of the group of patient before CONSOL is implemented. The investigators will match the 2 groups on time period (e.g., CONSOL group recruited in 6-month period with pre-CONSOL group in the 6 months prior CONSOL.
  Vital sign measured is heart rate. Abnormal vital sign cutoffs are listed below:
  Heart Rate (beats/minute) 1-4 years old < 60 or >120 5-12 years old <60 or >110 13-18 years old <60 or >100
Change in respiratory rate with CONSOL compared to pre-CONSOL implementation | During the intervention (vital sign monitoring using the Garmin Venu 3)
  The investigators will implement CONSOL and record the abnormal vital signs indicative of clinically meaningful events in the CONSOL group. The investigators will then compare the number of abnormal vital signs detected in the CONSOL group to that of the group of patient before CONSOL is implemented. The investigators will match the 2 groups on time period (e.g., CONSOL group recruited in 6-month period with pre-CONSOL group in the 6 months prior CONSOL.
  Vital sign measured respiratory rate. Abnormal vital sign cutoffs are listed below:
  Respiratory Rate (breaths/minute) 1-4 years old <20 or >30 5-12 years old <16 or >20 13-18 years old <12 or >16
Change in SPO2 with CONSOL compared to pre-CONSOL implementation | During the intervention (vital sign monitoring using the Garmin Venu 3)
  The investigators will implement CONSOL and record the abnormal vital signs indicative of clinically meaningful events in the CONSOL group. The investigators will then compare the number of abnormal vital signs detected in the CONSOL group to that of the group of patient before CONSOL is implemented. The investigators will match the 2 groups on time period (e.g., CONSOL group recruited in 6-month period with pre-CONSOL group in the 6 months prior CONSOL.
  Vital sign measured SPO2. Abnormal vital sign cutoffs are listed below:
  SPO2<92%

SECONDARY OUTCOMES:
Change in time to detection of abnormal heart rate using CONSOL | During the intervention (vital sign monitoring using the Garmin Venu 3)
  Change in time to detection of abnormal heart rate (HR) will be estimated by assessing detection of abnormal HR in intervals of 15 minutes up to 6 hours (usual care intervals of manual VS measurement). Since CONSOL will be implemented in addition to usual care manual HR measurement, abnormal HR detected by CONSOL can be compared to abnormal HR detected by manual measurement at each interval.
  Abnormal heart rate cutoffs are listed below:
  Heart Rate (beats/minute) 1-4 years old < 60 or >120 5-12 years old <60 or >110 13-18 years old <60 or >100
Change in time to detection of abnormal SPO2 using CONSOL | During the intervention (vital sign monitoring using the Garmin Venu 3)
  Change in time to detection of abnormal SPO2 will be estimated by assessing detection of abnormal SPO2 in intervals of 15 minutes up to 6 hours (usual care intervals of manual VS measurement). Since CONSOL will be implemented in addition to usual care manual SPO2 measurement, abnormal SPO2 detected by CONSOL can be compared to abnormal SPO2 detected by manual measurement at each interval.
  Abnormal SPO2, cutoffs are listed below:
  SpO2 (%) <92%
Change in time to detection of abnormal respiratory rate using CONSOL | During the intervention (vital sign monitoring using the Garmin Venu 3)
  Change in time to detection of abnormal respiratory rate (RR) will be estimated by assessing detection of abnormal RR in intervals of 15 minutes up to 6 hours (usual care intervals of manual RR measurement). Since CONSOL will be implemented in addition to usual care manual RR measurement, abnormal RR detected by CONSOL can be compared to abnormal RR detected by manual measurement at each interval.
  Abnormal respiratory rate cutoffs are listed below:
  Respiratory Rate (breaths/minute) 1-4 years old <20 or >30 5-12 years old <16 or >20 13-18 years old <12 or >16

OTHER OUTCOMES:
Exploratory outcome: Investigation of the dynamic heart rate patterns associated with clinical deterioration and rescue interventions | During the intervention (vital sign monitoring using the Garmin Venu 3)
  The dynamic VS patterns associated with clinical deterioration and rescue interventions will be examined only for patients who experienced a rescue intervention. Vital signs measured is heart rate. Rescue interventions are defined as actions taken to stabilize a patient with quickly deteriorating physiological status.
Exploratory outcome: Investigation of the dynamic SPO2 patterns associated with clinical deterioration and rescue interventions | During the intervention (vital sign monitoring using the Garmin Venu 3)
  The dynamic VS patterns associated with clinical deterioration and rescue interventions will be examined only for patients who experienced a rescue intervention. Vital signs measured is SPO2. Rescue interventions are defined as actions taken to stabilize a patient with quickly deteriorating physiological status.
Exploratory outcome: Investigation of the dynamic skin temperature patterns associated with clinical deterioration and rescue interventions | During the intervention (vital sign monitoring using the Garmin Venu 3)
  The dynamic VS patterns associated with clinical deterioration and rescue interventions will be examined only for patients who experienced a rescue intervention. Vital signs measured is skin temperature. Rescue interventions are defined as actions taken to stabilize a patient with quickly deteriorating physiological status.
Exploratory outcome: Investigation of the dynamic respiratory rate patterns associated with clinical deterioration and rescue interventions | During the intervention (vital sign monitoring using the Garmin Venu 3)
  The dynamic VS patterns associated with clinical deterioration and rescue interventions will be examined only for patients who experienced a rescue intervention. Vital signs measured is respiratory rate. Rescue interventions are defined as actions taken to stabilize a patient with quickly deteriorating physiological status.

IPD SHARING:
Plan to Share IPD: No
IPDs are considered PHI and can only be shared in a de-identified form. We have plans to share these de-identified data on ICPSR as per the Data Management and Sharing plan required by NIH